CLINICAL TRIAL: NCT02121964
Title: Anterior Capsulectomy Versus Capsulotomy With Repair in Direct Anterior Total Hip Arthroplasty
Brief Title: Capsulectomy vs Capsulotomy With Repair in Direct Anterior Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas L Bradbury, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00054340
Record Dates: First submitted 2014-04-14; First posted 2014-04-24 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Hip Arthrosis; Osteoarthritis; Arthritis
Keywords: unilateral primary total hip arthroplasty; bilateral primary total hip arthroplasty; Arthritis; Orthopedic Disorders; Orthopedics; Surgery,; Orthopedic; arthroplasty; hip; osteoarthritis; capsulectomy; capsulotomy
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Arthritis; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsulectomy (Other): Capsulectomy in Direct Anterior Total Hip Arthroplasty
  Interventions: Procedure: Capsulectomy in Direct Anterior Total Hip Arthroplasty
- Capsulotomy (Other): Capsulotomy in Direct Anterior Total Hip Arthroplasty
  Interventions: Procedure: Capsulotomy in Direct Anterior Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Capsulectomy in Direct Anterior Total Hip Arthroplasty — Surgical intervention in which the surgeon will perform anterior capsulectomy during total hip arthroplasty.
  Arms: Capsulectomy
Procedure: Capsulotomy in Direct Anterior Total Hip Arthroplasty — Surgical intervention in which the surgeon will perform anterior capsulotomy during total hip arthroplasty. Surgeon will repair the joint capsule.
  Arms: Capsulotomy

SUMMARY:
In this prospective, randomized study, investigators will look at the outcome of total hip arthroplasty through the anterior approach in regard to the surgical treatment of the anterior hip capsule. At this time, there are 2 different techniques: one is excising this capsule and the second one is cutting the capsule and repairing it at the end of the procedure. The investigators set out to determine whether incising or repairing the capsule will benefit the patients in terms of postoperative pain level, range of motion of the hip joint, joint stability, surgical time and blood loss. Both preserving and excising the joint capsule are accepted techniques in performing total hip arthroplasty. The Investigators hypothesize that capsulectomy may allow for reduction in operative time, provide superior surgical exposure, and increased range of motion after surgery. The influence on post operative pain and dislocation rate is unknown.

DETAILED DESCRIPTION:
Utilization of the direct anterior approach for total hip arthroplasty (THA) has increased over the last ten years. The approach, as described by Keggi et al, superficially utilizes the internervous muscle plane between the tensor fascia lata and the sartorius and deeply between the rectus and gluteus medius (1). Performing this muscle sparing rather than muscle splitting approach has several purported benefits. The clinical reports of this surgical approach have documented low dislocation rates (2, 3), excellent cup position (4) improved outcome scores (5), less muscle damage (6, 7) and improved gait mechanics (8). The preservation and repair of the anterior hip capsule (iliofemoral and pubofemoral ligaments) has been recommended by some authors, while anterior capsulectomy has been described by other authors without a reported increase in dislocation rate. In contrast, the higher risk of posterior dislocation using the posterior approach improved significantly after repair of the capsule (9, 10). There are no studies to date that have investigated outcome scores based on capsular repair versus capsulectomy for the THA direct anterior approach. The effects of anterior capsular repair versus capsulectomy are unknown with regards to anterior hip pain, range of motion, and surgical recovery. We hypothesize that capsulectomy may allow for reduction in operative time, provide superior surgical exposure, and increased range of motion after surgery. The influence on post operative pain and dislocation rate is unknown.

In this prospective, randomized clinical study investigators will compare operative time, blood loss, postoperative pain, range of motion, strength, and adverse events using two different surgical techniques (anterior capsular repair versus anterior capsulectomy) during direct anterior total hip arthroplasty. Patients will be randomized at their screening visit to one of two groups (anterior capsule repair or anterior capsulectomy), and they will be blinded for the group assignment. The surgical procedures will be performed according to the surgeon's routine standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral or bilateral primary total hip arthroplasty
* Direct anterior surgical approach
* Osteoarthritis diagnosis
* 18 years of age or older

Exclusion Criteria:

* Revision hip arthroplasty
* Avascular necrosis of the hip
* Rheumatoid arthritis of the hip
* Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Range of Motion- Resisted Hip Flexion Strength | Follow Up Visit (Up to six months)
  Measurement will be recorded taken with patient in the seated position with the hip flexed to 90 degrees. Strength will be measured when resistance is applied to the knee as the patient brings the leg up. The following scale will be used (each may be +/-, i.e. 5+):
  * 5 = NORMAL - the patient is able to actively move through the full available range of motion (ROM) against gravity and against maximal resistance
  * 4 = GOOD - the patient is able to actively move through the full available ROM against gravity and against moderate resistance
  * 3 = MODERATE - the patient is able to actively move through greater than one half the available ROM against gravity and against moderate resistance
  * 2 = POOR - the patient is unable to actively flex hip against gravity
  * 1 = BAD - the patient is unable to flex muscle properly
Change in Range of Motion - Maximum Hip Flexion | Screening Visit, Follow-up visit (Up to six months)
  This angle will be measured with the patient in the supine position utilizing a goniometer (recorded in degrees). Patients will flex the hip by bringing their leg as close to their trunk as possible with their knee bent. The angle between the trunk and leg will be recorded
Change in Range of Motion - Maximum Hip Extension | Screening Visit, Follow Up Visit (Up to six months)
  This angle will be measured with the patient in the prone position utilizing a goniometer. The patient will raise the lower leg to the limit of extension. The angle between the leg and table is recorded.
Change in Range of Motion - Evidence of Flexion Contraction (Thomas Test) | Screening Visit, Follow Up Visit (Up to six months)
  This angle will be measured with the patient lying in the supine position. Patient will bring opposite knee to the chest, while the other leg remains extended. The angle between the extended leg and the table is recorded.
Change in Pain Score with Resisted Hip Flexion | Screening Visit, Follow Up Visit (Up to six months)
  Measured using the Pain Assessment scale (PAS) of 0-10 (0 being no pain; 10 being worst imaginable pain).

SECONDARY OUTCOMES:
Change in Hip Disability and Osteoarthritis Outcome Score | Screening Visit, Follow Up Visit (Up to six months)
  Hip disability and osteoarthritis outcome survey (HOOS) administered to patients.
Surgical Time | Inpatient Surgery Visit (Day 0)
  This will be measured from the time of incision to the time the dressing is applied (per registered nurse (RN) operating room record).
Transfusion Rate by Percent Hemoglobin Drop | Inpatient Surgery Visit (Day 0)
  This will be recorded by review of inpatient medical records. Percent hemoglobin drop will be measured by comparing the preoperative hemoglobin to the inpatient nadir hemoglobin.
Number of Adverse Events | Duration of study (Up to six months)
  Patients will be assessed for complications that occur as a result of THA. These will be assessed at the standard of care intervals (6 week and 6 month follow-up visits). Any change in stem position including subsidence and radiolucencies will be reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Bradbury, M.D., Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keggi KJ, Huo MH, Zatorski LE. Anterior approach to total hip replacement: surgical technique and clinical results of our first one thousand cases using non-cemented prostheses. Yale J Biol Med. 1993 May-Jun;66(3):243-56. PMID 8209560
- [Background] Matta JM, Shahrdar C, Ferguson T. Single-incision anterior approach for total hip arthroplasty on an orthopaedic table. Clin Orthop Relat Res. 2005 Dec;441:115-24. doi: 10.1097/01.blo.0000194309.70518.cb. PMID 16330993
- [Background] Restrepo C, Mortazavi SM, Brothers J, Parvizi J, Rothman RH. Hip dislocation: are hip precautions necessary in anterior approaches? Clin Orthop Relat Res. 2011 Feb;469(2):417-22. doi: 10.1007/s11999-010-1668-y. PMID 21076896
- [Background] Masonis J, Thompson C, Odum S. Safe and accurate: learning the direct anterior total hip arthroplasty. Orthopedics. 2008 Dec;31(12 Suppl 2):orthosupersite.com/view.asp?rID=37187. PMID 19298019
- [Background] Restrepo C, Parvizi J, Pour AE, Hozack WJ. Prospective randomized study of two surgical approaches for total hip arthroplasty. J Arthroplasty. 2010 Aug;25(5):671-9.e1. doi: 10.1016/j.arth.2010.02.002. Epub 2010 Apr 8. PMID 20378307
- [Background] Bremer AK, Kalberer F, Pfirrmann CW, Dora C. Soft-tissue changes in hip abductor muscles and tendons after total hip replacement: comparison between the direct anterior and the transgluteal approaches. J Bone Joint Surg Br. 2011 Jul;93(7):886-9. doi: 10.1302/0301-620X.93B7.25058. PMID 21705558
- [Background] Meneghini RM, Pagnano MW, Trousdale RT, Hozack WJ. Muscle damage during MIS total hip arthroplasty: Smith-Petersen versus posterior approach. Clin Orthop Relat Res. 2006 Dec;453:293-8. doi: 10.1097/01.blo.0000238859.46615.34. PMID 17006366
- [Background] Mayr E, Nogler M, Benedetti MG, Kessler O, Reinthaler A, Krismer M, Leardini A. A prospective randomized assessment of earlier functional recovery in THA patients treated by minimally invasive direct anterior approach: a gait analysis study. Clin Biomech (Bristol). 2009 Dec;24(10):812-8. doi: 10.1016/j.clinbiomech.2009.07.010. Epub 2009 Aug 21. PMID 19699566
- [Background] Pellicci PM, Bostrom M, Poss R. Posterior approach to total hip replacement using enhanced posterior soft tissue repair. Clin Orthop Relat Res. 1998 Oct;(355):224-8. doi: 10.1097/00003086-199810000-00023. PMID 9917607
- [Background] Weeden SH, Paprosky WG, Bowling JW. The early dislocation rate in primary total hip arthroplasty following the posterior approach with posterior soft-tissue repair. J Arthroplasty. 2003 Sep;18(6):709-13. doi: 10.1016/s0883-5403(03)00254-7. PMID 14513442
- [Derived] Schwartz AM, Goel RK, Sweeney AP, Bradbury TL Jr. Capsular Management in Direct Anterior Total Hip Arthroplasty: A Randomized, Single-Blind, Controlled Trial. J Arthroplasty. 2021 Aug;36(8):2836-2842. doi: 10.1016/j.arth.2021.03.048. Epub 2021 Mar 26. PMID 33865648